CLINICAL TRIAL: NCT00276406
Title: Pyridostigmine in Diabetics With Constipation: Randomized, Placebo-controlled, Double-blind Trial
Brief Title: Use of Pyridostigmine for Constipation in Diabetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, MD, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-004037; UL1RR024150-01 (NIH); P01DK068055 (NIH)
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Results first posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Constipation; Diabetes Mellitus; Colonic Transit; Gastric Emptying
MeSH Terms: conditions — Constipation; Diabetes Mellitus | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyridostigmine (Experimental): Oral pyridostigmine, starting with 60 mg capsules three times per day (TID), increasing by 60 mg every third day (i.e., over 10 days) up to the maximum tolerated dose or 120 mg TID (a total of 360 mg per day). This dose was maintained for 7 days.
  Interventions: Drug: Pyridostigmine
- Placebo (Placebo Comparator): Placebo (sham) capsules, matching the appearance of the active drug comparator and taken TID.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyridostigmine — Pyridostigmine will be started at (60mg) tid, increased over 10 days to 120 mg tid, and maintained at that dose for 7 days.
  Other Names: Mestinon
  Arms: Pyridostigmine
Drug: Placebo — If subject is randomized to placebo, placebo pills will be started at (60mg) tid, increased over 10 days to 120 mg tid, and maintained at that dose for 7 days.
  Arms: Placebo

SUMMARY:
Doctors at Mayo Clinic are doing this study to learn if pyridostigmine, a drug, affects the speed at which food travels through the stomach, intestines and colon, and if pyridostigmine improves constipation symptoms in patients with diabetes. Pyridostigmine has been approved by the Food and Drug Administration (FDA) for routine clinical use, however, its use as proposed in this study is considered investigational.

DETAILED DESCRIPTION:
Chronic constipation in diabetes mellitus is associated with colonic motor dysfunction and is managed with laxatives. Cholinesterase inhibitors increase colonic motility. The study evaluated the effects of a cholinesterase inhibitor (pyridostigmine vs. placebo) on gastrointestinal and colonic transit and bowel function in diabetic patients with constipation.

After a 9-day baseline period, patients with diabetes mellitus and chronic constipation without defecatory disorder will be randomized to oral placebo or pyridostigmine, starting with 60 mg three times a day, increasing by 60 mg every third day up to the maximum tolerated dose of 120 mg three times a day; this dose will be maintained for 7 days. Gastrointestinal and colonic transit (assessed by scintigraphy) and bowel function will be evaluated at baseline and the final 3 and 7 days of treatment, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetes mellitus (Type I or type II), diagnosed by a physician.
* On medical treatment for diabetes (oral medication or injected insulin) for at least one year
* Symptomatic constipation at least 25% of the time in the past year (Rome II criteria for functional constipation)
* 18-70 years of age
* Colonoscopy negative for obstructive lesions, cancer, or inflammatory bowel disease (IBS) within the last 8 years if 50 years of age or older
* Able to provide written informed consent before participating in trial
* Able to communicate adequately with the Investigator and to comply with the requirements for the entire study

Exclusion Criteria:

* History of pelvic floor dysfunction (other functional GI disorders, eg IBS, non-ulcer dyspepsia are acceptable); Specifically, patients will be excluded if they have at least 2 of the following 3 criteria:

  * History of digital evacuation of the rectum or pressure on the posterior aspect of the vagina or perineum to facilitate defecation
  * Examination findings suggestive of puborectalis spasm or anismus, on assessment by an experienced gastroenterologist with expertise in this field; i.e. high anal sphincter tone at rest, failure of perineal descent by >1cm on straining, and tenderness or paradoxical contraction of the puborectalis on digital examination
  * Requirement of > 200g to expel a rectal balloon during voluntary straining
* Abdominal surgery other than appendectomy, cholecystectomy, hysterectomy, tubal ligation, or inguinal hernia repair
* Suspected or known gastrointestinal or genitourinary obstruction
* Uncontrolled hypertension (defined as > 150/90 at rest)
* Known cardiac arrhythmia or ECG abnormalities, i.e. cardiac conduction disturbances (2nd or 3rd degree atrioventricular (AV) block, prolonged corrected QT interval (QTc)(> 460 msec) or bradycardia (< 45 beats/minute))
* Renal insufficiency with serum creatinine greater than 2 mg/dl based on a reading from the previous 6 months
* Asthma or chronic obstructive pulmonary disease requiring systemic steroids in the previous 3 years (inhaled steroids acceptable)
* Current use of narcotics, gut prokinetic drugs (eg metoclopramide, domperidone, tegaserod, senekot), anticholinergic medication (eg. Hyoscyamine, belladonna), antidiarrheals (Imodium, Lomotil), or laxatives other than fiber supplements, docusate, or glycerin suppositories. Patients on any of these restricted medications must cease use at least 48 hours before starting and for the duration of both study phases. No rescue laxatives will be permitted within 7 days of transit testing
* Patients who have taken any investigational medications within the past 30 days
* Known intolerance or allergy to eggs
* Pregnant or breast-feeding females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E. Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Bharucha AE, Low P, Camilleri M, Veil E, Burton D, Kudva Y, Shah P, Gehrking T, Zinsmeister AR. A randomised controlled study of the effect of cholinesterase inhibition on colon function in patients with diabetes mellitus and constipation. Gut. 2013 May;62(5):708-15. doi: 10.1136/gutjnl-2012-302483. Epub 2012 Jun 7. PMID 22677718

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Mayo Clinic in Rochester, Minnesota and the study was conducted at between May 2006 and October 2010.
Pre-assignment Details: 68 patients were assessed for eligibility. 24 were ineligible. 13 were eligible but declined to participate in the study. One patient consented but was withdrawn because of severe hyperglycemia during the baseline period. 30 were enrolled and completed all study procedures.
Period: Overall Study
Arm/Group | Pyridostigmine | Placebo
Started | 16 | 14
Completed | 16 (14 of 16 subjects tolerated 360mg daily, while 2 of 16 tolerated 180mg daily.) | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pyridostigmine | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 48.5 (11.4) | 52.1 (11.3) | 50.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 3 | 5 | 8
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30
Body Mass Index [Mean (Standard Deviation); unit: kilograms/meter^2] — Body Mass Index (BMI) is a health index for comparing weight to height. BMI is a person's weight in kilograms (kg) divided by his or her height in meters squared. The body mass index is an indication if a person is at a suitable weight for his height on an approximation of body fat. A body mass index of under 20 is considered to be underweight, while a body mass index between 20 to 25 is considered healthy. A body mass index in the range of 25 to 30 is regarded as overweight. A body mass index over 30 is regarded as obese.
  kilograms/meter^2 | 27.9 (4.4) | 31.6 (6.0) | 29.7 (5.5)
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage] — Hemoglobin A1c (HgA1c) or glycolated hemoglobin is a laboratory test of blood which provides a measure the average blood glucose (sugar) levels for the prior 3 month period.
  Percentage | 8.1 (1.7) | 7.7 (1.2) | 7.9 (0.3)
Subjects with diabetic retinopathy [Number; unit: Participants] — Diabetic retinopathy is a condition of the eye caused by diabetes, caused by abnormal blood vessel growth, which invades the retina and can cause reduced vision and blindness.
  Note: because not all subjects had retinopathy, the number of subjects with retinopathy in each arm will not match the overall number of subjects enrolled in each arm.
  Participants | 9 | 7 | 16
Geometric Center (GC) of Colonic transit [Mean (Standard Deviation); unit: Units on a scale] — The scintigraphic method is used to measure movement of large intestine contents. A radio-labeled isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule taken by mouth with a meal. Abdominal anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
  Units on a scale
    Geometric Center of Colonic Transit at 24 hr (GC24 | 1.96 (0.71) | 1.98 (0.62) | 1.97 (0.66)
    Geometric Center of Colonic Transit at 48 hr (GC48 | 2.92 (0.89) | 2.97 (1.00) | 2.94 (0.93)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Geometric Center at 24 Hours (GC24) Measured by Scintigraphy
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images of the abdomen are taken hourly for the first 6 hours after the radio-labeled meal, then at 8, 24 and 48 hours. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool. GC24 is the measurement taken at 24 hours after the radio-labeled meal.
Time Frame: Baseline period (days 7-9 ), Treatment period (days 14-17)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
units on a scale
  Baseline | 1.96 (0.18) | 1.98 (0.17)
  Treatment | 2.45 (0.20) | 1.84 (0.16)
Statistical Analysis 1: Comparison: Pyridostigmine vs Placebo; Analysis was adjusted for BMI and baseline values and incorporated Bonferroni corrections; Test type: Superiority or Other; p < 0.01, ANCOVA

2. Primary Outcome: Ascending Colon Emptying Half-time (AC t1/2) Measured in Hours
Description: Calculated by linear interpolation of values on the AC emptying curve.
Time Frame: Baseline period (days 7-9 ), Treatment period (days 14-17)
Measure: Mean (Standard Error); unit: hours
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
hours
  Baseline | 16.73 (2.30) | 20.59 (3.29)
  Treatment | 10.44 (1.40) | 18.77 (3.23)

3. Secondary Outcome: Gastric Emptying Half-time (GE t1/2)
Description: The measure of time for 50 percent of a radio-labeled meal to empty from the stomach.
Time Frame: Baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
minutes
  Baseline | 142 (19) | 141 (12)
  Treatment | 122 (13) | 121 (13.42)

4. Secondary Outcome: Colonic Filling at 6 Hours
Description: The proportion of a radio-labeled meal in the colon at 6 hours (identifiable by radio-labelled tracer to capsule eaten with meal), measured by scintigraphy. This is an indirect measurement of small-bowel transit time.
Time Frame: Baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: percentage of meal
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
percentage of meal
  Baseline | 37 (9) | 41 (10)
  Treatment | 53 (7) | 48 (9)

5. Secondary Outcome: Colonic Geometric Center at 48 Hours (GC48) as Measured by Scintigraphy
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly for the first 6 hours after the radio-labeled meal, then at 8, 24 and 48 hours. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool. GC48 is the measurement taken at 48 hours after the radio-labeled meal.
Time Frame: Baseline period (days 7-9 ), Treatment period (days 14-17)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
units on a scale
  Baseline | 2.92 (0.22) | 2.97 (0.27)
  Treatment | 3.59 (0.25) | 3.26 (0.27)
Statistical Analysis 1: Comparison: Pyridostigmine vs Placebo; Analysis was adjusted for BMI and baseline values and incorporated Bonferroni corrections; Test type: Superiority or Other; p = 0.096, ANCOVA

6. Secondary Outcome: Stool Frequency Per Day
Description: During 9 days of the baseline period and during 17 days of the treatment period, subjects used a daily diary to record the number of times per day they had a bowel movement. Only the 7 days of highest treatment dose will be used for comparison purposes.
Time Frame: Daily during baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: Number of bowel movements
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
Number of bowel movements
  Baseline | 0.95 (0.2) | 1.2 (0.2)
  Treatment | 1.5 (0.2) | 1.4 (0.2)
Statistical Analysis 1: Comparison: Pyridostigmine vs Placebo; Test type: Superiority or Other; p = 0.02, ANCOVA

7. Secondary Outcome: Stool Form/Consistency
Description: During 9 days of the baseline period and during 17 days of the treatment period, subjects used a daily diary to record a description of stool consistency according to the Bristol Stool Form Scale (ranging from 1 (hard lumps) to 7 (watery)). The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: Daily during baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
units on a scale
  Baseline | 2.5 (0.3) | 2.8 (0.5)
  Treatment | 3.4 (0.2) | 2.6 (0.4)
Statistical Analysis 1: Comparison: Pyridostigmine vs Placebo; Bowel diaries were analyzed by computing the mean scores for the 9-day baseline period and separately for the last 7 days of the treatment period (i.e., when the pyridostigmine dose was stable in each subject.) Individual subject treatment period mean bowel function scores were then compared using a similar ANCOVA model, with the corresponding individual subject baseline mean bowel function score and gender as covariates; Test type: Superiority or Other; p = 0.005, ANCOVA

8. Secondary Outcome: Stool Ease of Passage
Description: During 9 days of the baseline period and during 17 days of the treatment period, subjects used a daily diary to record a description of stool ease of passage of stool, according to the Bristol Stool Form Scale (ranging from 1 (manual disimpaction) to 7 (incontinence)). Only the 7 days at highest treatment dose will be used for comparison purposes.
Time Frame: Daily during baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
units on a scale
  Baseline | 3.5 (0.2) | 3.6 (0.2)
  Treatment | 3.8 (0.5) | 3.5 (0.2)
Statistical Analysis 1: Comparison: Pyridostigmine vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p < 0.04, ANCOVA

9. Secondary Outcome: Sense of Completely Emptying Bowels
Description: During 9 days of the baseline period and during 17 days of the treatment period, subjects used a daily diary to record whether or not they felt they had completely emptied their bowels(1= Yes; 0= No). Only the 7 days of highest treatment dose will be used for comparison purposes.
Time Frame: Daily during baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: percentage of bowel movements
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
percentage of bowel movements
  Baseline | 86 (6) | 74 (8)
  Treatment | 73 (8) | 66 (8)

10. Secondary Outcome: Stool Frequency Per Week
Description: During 9 days of the baseline period and during 17 days of the treatment period, subjects used a daily diary to record the number of times per day they had a bowel movement. Complete spontaneous bowel movements per week are reported. Only the 7 days of highest treatment dose will be used for comparison purposes.
Time Frame: Daily during baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: Number complete bowel movements per week
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
Number complete bowel movements per week
  Baseline | 2.1 (0.9) | 2.1 (0.8)
  Treatment | 4.0 (1.2) | 3.1 (0.9)

11. Secondary Outcome: Heart Rate Before and After Treatment
Description: Heart rate is the number of beats per minute, as recording on an Electrocardiogram (ECG).
Time Frame: Baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
beats per minute
  Baseline | 74 (3) | 76 (4)
  Treatment | 66 (2) | 75 (3)

12. Secondary Outcome: QTc Interval Before and After Treatment
Description: The corrected QT interval (QTc) is a measurement of time (seconds) between the Q and T waves of an heart beat as recorded during an Electrocardiogram (ECG).
Time Frame: Baseline period (9 days), Treatment period (7 days)
Measure: Mean (Standard Error); unit: Milliseconds
Arm/Group | Pyridostigmine | Placebo
Number analyzed (Participants) | 16 | 14
Milliseconds
  Baseline | 428 (6) | 420 (8)
  Treatment | 415 (18) | 421 (4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the baseline (9 days) and treatment (7 days) periods. Events occuring in more than one subject are tabulated by treatment arm.
Arm/Group | Pyridostigmine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 11/16 | 5/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pyridostigmine (N=16) | Placebo (N=14)
Increased salivation and/or sweating (General disorders) | 3 (3) | 2 (2)
Muscle twitching (Nervous system disorders) | 3 (3) | 1 (1)
Abdominal discomfort, nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Fatigue, lightheadedness (General disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bluish discoloration of urine (Renal and urinary disorders) | 1 (1) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No